CLINICAL TRIAL: NCT07304648
Title: The Role of End-Tidal Carbon Dioxide Changes During Passive Leg Raising in Predicting Fluid Responsiveness for Mechanically Ventilated Patients in the Intensive Care Unit: A Prospective Observational Study
Brief Title: Role of End-Tidal CO2 During Passive Leg Raising to Predict Fluid Responsiveness in ICU
Status: Not yet recruiting | Type: Observational
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ahmet Salih Tüzen, MD, Medical Doctor, Izmir Katip Celebi University
Other Study IDs: 2025-SAEK-0807
Record Dates: First submitted 2025-12-13; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Circulatory Failure; Critical Illness; Hypovolemia
Keywords: Fluid Responsiveness; Passive Leg Raising; End-Tidal CO2; Mini Fluid Challenge; Mechanical Ventilation; Intensive Care
MeSH Terms: conditions — Shock; Critical Illness; Hypovolemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fluid Responders: Patients who demonstrate a significant hemodynamic improvement following the Mini Fluid Challenge (MFC. Defined as an increase in Left Ventricular Outflow Tract Velocity Time Integral (LVOT-VTI) of >10%. If VTI unavailable, increase in Systolic Arterial Pressure > 4%, Pulse Pressure variation decrease > 2%, or Mean Arterial Pressure increase > 15%.
- Fluid Non-Responders: Patients who do not demonstrate a significant hemodynamic improvement following the Mini Fluid Challenge (MFC). Defined as an increase in LVOT-VTI of < 10% (or failure to meet the alternative blood pressure criteria).

SUMMARY:
This prospective observational study evaluates whether monitoring changes in exhaled carbon dioxide (End-Tidal CO2 or EtCO2) during a "Passive Leg Raising" (PLR) test can reliably predict fluid responsiveness in critically ill patients.

In the Intensive Care Unit (ICU), fluid management is a critical balance; while fluid is necessary for tissue perfusion, overload can lead to severe complications. Traditional static measurements (like central venous pressure) are often unreliable for guiding therapy. Dynamic tests like PLR are preferred as they simulate a fluid bolus reversibly by shifting blood from the legs to the heart.

Researchers will observe mechanically ventilated patients planned for fluid resuscitation. The study compares the accuracy of non-invasive EtCO2 changes during PLR against a reference standard "Mini Fluid Challenge" (100 mL fluid administration). Fluid responsiveness will be confirmed using echocardiographic measurements (LVOT-VTI) or arterial pressure changes. The goal is to validate EtCO2 as a practical, real-time tool for safe fluid management.

DETAILED DESCRIPTION:
Fluid management is the cornerstone of hemodynamic stabilization in ICU patients with circulatory failure. However, distinguishing between patients who will benefit from fluid (responders) and those who will not is vital to prevent the high mortality associated with inappropriate fluid administration.Static parameters (e.g., CVP, MAP) fail to reliably predict fluid responsiveness. Dynamic parameters are superior but have limitations, such as dependence on regular heart rhythm and specific ventilation settings. Consequently, interest has shifted toward non-invasive surrogates for cardiac output, such as End-Tidal CO2 (EtCO2), which tracks pulmonary blood flow changes under constant ventilation. This study investigates whether Delta EtCO2 during a PLR maneuver can accurately predict the response to a fluid challenge. The primary objective is to determine the diagnostic accuracy of Delta EtCO2 during PLR. Its predictive value will be validated against the hemodynamic response to a Mini Fluid Challenge (MFC), serving as the reference method. This prospective, single-center, observational cohort study includes adult patients in the ICU receiving mechanical ventilation who require fluid resuscitation.

Passive Leg Raising (PLR) Test: The patient starts in a semi-recumbent position (45°). They are then moved to a supine position with legs raised to 45° without manual handling to avoid sympathetic stimulation. This auto-transfuses blood from the lower body to the central circulation, increasing preload.

Mini Fluid Challenge (MFC): Following PLR, 100 mL of crystalloid fluid is infused intravenously over approximately 1 minute.

Definition of Fluid Responsiveness (Reference Standard): An increase in Left Ventricular Outflow Tract Velocity Time Integral (LVOT-VTI) of >10% on echocardiography. If cardiac output/VTI cannot be assessed, responsiveness is defined as a Systolic Arterial Pressure increase of > 4%, a Pulse Pressure variation decrease of > 2%, or a Mean Arterial Pressure increase of > 15%.

The sample size was calculated using G*Power 3.1 software based on a pilot study of 6 patients. In the pilot study, Delta EtCO2 values were found to be 3.5±2.1 mmHg in the fluid responder group and 2.1±1.1 mmHg in the non-responder group. Based on these findings, with an effect size (Cohen's d) of 0.72, an alpha error level of 0.05, and a targeted power (1-beta) of 0.80, the required sample size was calculated. Accounting for a potential 10% attrition rate, the study is planned to be conducted with a total of 68 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older.
* Patients who have been followed in the intensive care unit (ICU) with mechanical ventilation support for at least 24 hours.
* Patients for whom a mini fluid challenge (MFC) is clinically planned by the intensive care team.
* Patients for whom informed consent has been obtained from first-degree relatives or a legal representative.

Exclusion Criteria:

* Patients younger than 18 years of age.
* Pregnant patients.
* Patients without consent from first-degree relatives or a legal representative.
* Patients with known deep vein thrombosis (DVT) in the leg veins (risk of embolism during leg raising).
* Patients with pathologies that may cause increased intracranial pressure (e.g., intracranial mass, hemorrhage).
* Patients with uncontrolled hypertension.
* Patients with severe cardiac disease (e.g., right heart failure, pulmonary hypertension, advanced valvular pathology).
* Patients with carbon dioxide (CO2) retention.
* Patients who have undergone hip surgery or hip replacement surgery where Passive Leg Raising (PLR) cannot be performed.
* Patients with spontaneous breathing.
* Patients with a probability of high intra-abdominal pressure.
* Patients who cannot lie in a supine position.
* Patients with current peripheral oxygen saturation (SpO2) < 88%.
* Patients on mechanical ventilation requiring pressure support > 16 mmHg or PEEP > 10 mmHg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients (aged 18 years or older) admitted to the Intensive Care Unit (ICU) of a university hospital. Eligible participants are those who have been receiving mechanical ventilation support for at least 24 hours and have been identified by the primary intensive care team as requiring a fluid responsiveness assessment via a mini fluid challenge. The cohort includes patients with circulatory failure or suspected hypovolemia where fluid resuscitation is clinically indicated. Patients with contraindications to passive leg raising (e.g., intracranial hypertension, deep vein thrombosis), spontaneous breathing, or severe cardiac valve pathologies are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in End-Tidal Carbon Dioxide (Delta EtCO2) during Passive Leg Raising (PLR) | Measured between 60 to 90 seconds after the position change.
  The absolute difference in End-Tidal CO2 (EtCO2) levels will be calculated between the baseline measurement (T0, patient semi-recumbent at 45°) and the measurement taken during the Passive Leg Raising test (T1, patient supine with legs raised to 45°). The diagnostic accuracy of this Delta EtCO2 will be evaluated by comparing it against the patient's fluid responsiveness status (Responder vs. Non-Responder) determined by the subsequent Mini Fluid Challenge.

SECONDARY OUTCOMES:
Change in Arterial Blood Pressures (SAP, DAP, MAP) | Measured between 60 to 90 seconds after the position change.
  Systolic (SAP), Diastolic (DAP), and Mean Arterial Pressure (MAP) will be monitored at baseline (T0) and during the PLR maneuver (T1). The changes in these pressures will be compared between the fluid responder and non-responder groups.
Change in Heart Rate (Delta HR) | Measured between 60 to 90 seconds after the position change.
  Heart rate will be monitored at baseline (T0) and during the PLR maneuver (T1). The absolute change (Delta HR) will be compared between the fluid responder and non-responder groups.
Change in Pulse Pressure Variation (Delta PPV) | Measured between 60 to 90 seconds after the position change.
  Pulse Pressure Variation (PPV) will be monitored at baseline (T0) and during the PLR maneuver (T1). The change in PPV will be compared between the fluid responder and non-responder groups.
Change in Oxygen Saturation (Delta SO2) | Measured between 60 to 90 seconds after the position change.
  Oxygen Saturation (SO2) will be monitored at baseline (T0) and during the PLR maneuver (T1). The change will be compared between the fluid responder and non-responder groups.
Change in Vena Cava Inferior (VCI) Distensibility Index | Measured between 60 to 90 seconds after the position change.
  The VCI diameter will be measured using ultrasonography during inspiration and expiration at baseline (T0) and during the PLR maneuver (T1). The VCI distensibility index will be calculated and its change compared between the groups.
Change in Left Ventricular Outflow Tract Velocity Time Integral (LVOT-VTI) | Immediately following the 1-minute Mini Fluid Challenge.
  This is the reference standard used to classify patients. Following the Mini Fluid Challenge (100ml crystalloid over 1 min), the percentage change in LVOT-VTI is measured. An increase of >10% defines the patient as a "Fluid Responder".

CONTACTS AND LOCATIONS:
Overall Officials: Murat Aksun, M.D., Principal Investigator — Izmir Katip Celebi University Atatürk Training and Research Hospital
Locations (1):
- Izmir Katip Celebi University Atatürk Training and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
All data necessary to support the study protocol, including de-identified individual participant data (IPD) related to study protocol, and primary and secondary outcome measures, will be made available upon reasonable request from qualified researchers for academic purposes, in accordance with institutional and ethical guidelines.